CLINICAL TRIAL: NCT04485741
Title: Clinical Utility of Strados System in Periodically Recording Auscultation to Provide Replay Capability and Telemedicine Monitoring of Inpatients After Initial Clinical Assessment.
Brief Title: Strados System at Center of Excellence
Status: Completed | Type: Observational
Sponsor: Strados Labs, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: SL-RS-AEMC01
Record Dates: First submitted 2020-07-21; First posted 2020-07-24 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2023-01

CONDITIONS: Copd; Asthma; Covid19
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Asthma; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: RESP — The RESP device will be placed on the patient for periodic recording of auscultory sound.
  Other Names: Strados System

SUMMARY:
Listening to breath sounds with the stethoscope/auscultation is used by pulmonary physicians in conjunction with pulmonary function, signs and symptoms, oxygen saturation and diagnostic testing to admit, follow and discharge patients from hospital. Of these, only auscultation routinely ceases upon discharge from Hospital. Healthcare utilization statistics have shown that for more than a decade, readmission after discharge for an exacerbation of COPD or severe asthma (or chronic heart failure) remains a major problem. The Strados System has been designed to extend the range of lung sound recording both geographically and temporally to improve the standard of care when access to continuous monitoring has been replaced by periodic or no monitoring. The primary purpose of this study is to assess the clinical utility of the Strados System in enabling periodic recording and reviewing of breath sounds in patients with chronic respiratory diseases, either in the ICU, or in less continuously monitored settings, including after inpatient discharge.

ELIGIBILITY:
Inclusion Criteria:

Potential study participants will be recruited from within the Einstein Center of Excellence. Individuals who meet all of the following criteria are eligible for enrollment as study participants:

1. Males and females between the ages of 18-80:

   With documented physician-diagnosed COPD (chronic bronchitis dominant) or severe asthma, as defined either by the American Thoracic Society or the World Health Organization who are admitted for exacerbation, including those with active or suspected SARS-COV-2 infection

   OR

   Who are admitted with respiratory distress symptoms associated with SARS-COV-2 infection
2. Able to provide informed consent
3. Able to follow study procedures
4. Clinician assessment of the patient's current SARS-COV-2 status: negative or unlikely to be infected, RTPCR positive, or untested by clinically suspected
5. Accessible by telephone upon discharge

Exclusion Criteria:

Subjects who meet ANY of the following criteria are not eligible for enrollment:

1. Inability or unwillingness of the participant to give written informed consent
2. History of adverse reaction or allergy to Tegaderm
3. Unwillingness or inability to comply with study procedures
4. Scheduled for thoracic procedure
5. Inaccessible by telephone post-discharge

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who are admitted for exacerbation of chronic airway disease (COPD or severe asthma) or for respiratory distress symptoms associated with SARS-COV-2 infection for 1 to 3 weeks to ICU or specialty floor with access to telemedicine monitoring
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2020-09-23 (Actual); Primary Completion 2021-12-28 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Clinical utility as assessed by the PI | Periodic recording over 12 to 24 hours
  To assess the clinical utility of Strados Systems in enabling periodic recording and reviewing of lung breath sounds of inpatients with chronic respiratory diseases in ICU , and less continuously monitored settings.

SECONDARY OUTCOMES:
Clinical utility as assessed by other clinicians | Periodic recording over 12 to 24 hours
Correlation of RESP data with other measures of patient status. | Periodic recording over 12 to 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Albert Einstein Medical Center, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided